CLINICAL TRIAL: NCT00159549
Title: Long Term Effect of an Education and Training Program for Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMF 05/414
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Patient education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

INTERVENTIONS:
Behavioral: education and training program

SUMMARY:
A parallell group study comparing the effect of an education program with an education and training program for patients with COPD. 30 participants in each group. Participants self-select which group they wanted to be in. Main outcome is SGRQ (a HQoL for patients with COPD).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD (FEV1<75% of expected) who have the ability to conversation and active participation will be included.

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2000-01 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
St Geoprg Respiratory Questionnaire (SGRQ)

SECONDARY OUTCOMES:
COPD-Efficacy scale (Norwegian short version), Breathing Problems Questionnaire (BPQ), journal examinations, FVC, FEV1, six minutes walking test with registration of shortness of breath and pulseoxymetrical data.

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Steinsbekk, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Community Medicine and General Practice, Trondheim, Norway

REFERENCES:
- [Result] Lomundal BK, Steinsbekk A. Observational studies of a one year self-management program and a two year pulmonary rehabilitation program in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2007;2(4):617-24. PMID 18268936
- [Result] Steinsbekk A, Lomundal BK. Three-year follow-up after a two-year comprehensive pulmonary rehabilitation program. Chron Respir Dis. 2009;6(1):5-11. doi: 10.1177/1479972308098387. PMID 19176707